CLINICAL TRIAL: NCT02158975
Title: Open-label, Single-center Phase II Study of MLN9708 (Ixazomib) in Patients With Relapsed/Refractory Cutaneous and Peripheral T-cell Lymphomas
Brief Title: Open-label, Phase II Study of MLN9708 in Patients With Relapsed/Refractory Cutaneous and Peripheral T-cell Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2014.031; HUM00088647 (Other: University of Michigan)
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Lymphoma, T-Cell
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MLN9708 (Experimental): MLN9708 4mg by mouth weekly (days 1, 8, 15) every 28 days.
  Interventions: Drug: MLN9708

INTERVENTIONS:
Drug: MLN9708

SUMMARY:
Historically cutaneous and peripheral T-cell lymphomas have response rates of approximately 30% to standard chemotherapy regimens. We alternatively hypothesize that MLN9708 will be active in this disease and will improve best objective response.

We will also determine the extent to which MLN9708 inhibits GATA-3 (Trans-acting T-cell-specific transcription factor) expression, which is associated with poor prognosis, and whether GATA-3 expression represents a novel predictive biomarker for MLN9708 sensitivity.

DETAILED DESCRIPTION:
Up to 25 patients meeting the inclusion and exclusion criteria will be enrolled into this trial in two stages. All enrolled patients will be treated with MLN9708 4 mg PO weekly (days 1, 8, 15 every 28 days) until disease progression or unacceptable toxicity. In the initial stage of the study a total of 11 patients will be enrolled and treated with MLN9708. Should at least 4 patients exhibit a response (CR/CRu, PR), the second stage of 14 patients will open for enrollment. Efficacy will be assessed radiographically, by peripheral blood and bone marrow examination (when indicated), and physical exam every 8 weeks. Safety will be assessed by periodic physical exams, laboratory studies, and adverse events. All patients will have a follow-up visit 35 days (+/-7 days) following the last study drug treatment. Patients with accessible tumor tissue will be asked to undergo a biopsy for a fresh tissue sample for assessment of GATA-3 expression. Archived tissue samples from the initial diagnostic biopsy and the most recent lymphoma biopsy will be obtained in the event a fresh tumor biopsy cannot be obtained. Patients with GATA-3+ TCL and accessible tumor tissue will undergo a tumor biopsy at day 21 (+/- 7 days) of cycle 1. All baseline fresh or archived tissue will undergo central pathology review to confirm the diagnosis of TCL. The rationale for proteasome inhibition in T-cell lymphomas, based on the pre-clinical (and previous phase II) data, is compelling. Therefore, this phase II study will not be restricted to patients with GATA-3 expressing lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older at the time of enrollment.
* Voluntary written consent must be given.
* Female patients who are postmenopausal for at least 1 year before the screening visit, OR surgically sterile, OR agree to practice 2 effective methods of contraception, at the same time, through 90 days after the last dose of study drug, AND adhere to the guidelines of any treatment-specific pregnancy prevention program, OR agree to practice true abstinence.
* Male patients must agree to practice effective barrier contraception through 90 days after the last dose of study drug, OR adhere to the guidelines of any treatment-specific pregnancy prevention program, OR agree to practice true abstinence.
* Patients must have histologically proven T-cell lymphoma, including Peripheral T-cell lymphoma, Angioimmunoblastic T-cell lymphoma, Anaplastic large cell lymphoma (ALK positive), Anaplastic large cell lymphoma (ALK negative), Mycosis fungoides, Sezary syndrome.
* CTCL patients must have stage IIb-IV disease.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet count ≥ 75,000/mm3.
* Platelet transfusions are not allowed within 3 days before study enrollment.
* Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ to 3 x ULN.
* Creatinine clearance ≥30 mL/min.
* Documented disease progression after receiving at least one prior therapeutic regimen.

Exclusion Criteria:

* Female patients who are lactating or have a positive serum pregnancy test.
* Failure to have recovered (ie, less than or equal to Grade 1 toxicity) from the reversible effects of prior chemotherapy.
* Major surgery within 14 days of enrollment.
* Radiotherapy within 14 days of enrollment. If the field is small, 7 days will be considered a sufficient interval between treatment and administration of the MLN9708.
* Known central nervous system involvement.
* Infection requiring systemic intravenous antibiotic therapy or other serious infection within 7 days before study enrollment.
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
* Systemic treatment, within 14 days before the first dose of MLN9708, with strong inhibitors of CYP1A2, strong inhibitors of CYP3A or strong CYP3A inducers or use of Ginkgo biloba or St. John's wort.
* Ongoing or active systemic infection, active hepatitis B or C virus infection, or HIV positive.
* Any serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
* Known allergy to any of the study medications, their analogues, or excipients.
* Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of MLN9708 including difficulty swallowing.
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Patient has greater than or equal to Grade 3 peripheral neuropathy, or Grade 2 with pain on clinical examination during the screening period.
* Participation in other clinical trials with other investigational agents not included in this trial, within 21days of the start of this trial and throughout the duration of this trial.
* Prior allogeneic hematopoietic stem cell transplant.
* Prior autologous hematopoietic stem cell transplant within 90 days of study entry.
* Prior treatment with bortezomib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-09; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Wilcox, M.D., Ph.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- MLN9708: MLN9708 4mg by mouth weekly (days 1, 8, 15) every 28 days.
  MLN9708
Period: Overall Study
Arm/Group | MLN9708
Started | 13
Completed | 12
Not Completed | 1
Not completed — Did not complete 1 cycle nor > 1dose | 1

BASELINE CHARACTERISTICS:
Population: 12 analyzable patients
Arm/Group | MLN9708
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 70 [55 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
T-Cell Lymphoma Subtype [Count of Participants; unit: Participants]
  Cutaneous T-cell Lymphoma (CTCL) | 5
  Peripheral T-cell Lymphoma (PTCL) | 7

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The percentage of patients with an objective response rate will be determined. The overall response will be based on response in each compartment (skin, blood, lymph nodes and viscera) using a global composite scoring system. Objective response is considered (CR) Complete Response (Complete disappearance of all clinical evidence of disease), CRu (Complete Response Unconfirmed), or (PR) Partial Response (Regression of measurable disease).
Time Frame: Up to 24 months after initiation of study treatment
Population: 12 analyzable patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | MLN9708
Number analyzed (Participants) | 12
percentage of patients | 8 [1.5 to 35]

2. Secondary Outcome: Number Patients That Experience Adverse Events, Grades 3-5
Description: To assess the safety and tolerability of MLN9708, the number of patients experiencing Adverse Events (AEs) greater than or equal to grade 3 will be recorded.
Time Frame: 30 days after the last dose of study drug
Measure: Number; unit: participants
Arm/Group | MLN9708
Number analyzed (Participants) | 12
participants
  Anemia | 1
  Thrombocytopenia | 1
  Diarrhea | 1
  Mucocitis | 1
  Acute Kidney Injury | 1
  Atrial Fibrilation | 1
  Dyspnea | 1
  Hypercalcemia | 1
  Hyponatremia | 1
  Hypotension | 1
  Lymph Node Pain | 1
  Rash | 1
  Respiratory Failure | 1
  Supraventricular Tachycardia | 1
  Thromboembolic Event | 1

3. Secondary Outcome: Median Progression Free Survival Time
Description: Progression Free Survival (PFS) is defined as the time from study start until disease progression or death.
Time Frame: 24 months after initiation of study treatment
Population: 5 of the 12 patients withdrew prior to progression and therefore progression free survival was censored at their time of withdraw.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MLN9708
Number analyzed (Participants) | 12
months | 3.2 [1.6 to NA] — the upper limit was not reached

4. Secondary Outcome: Median Overall Survival Time
Description: Overall Survival (OS) is defined as the time from study start until death.
Time Frame: 24 months after initiation of study treatment
Population: Five patients died between start of treatment and database lock. Patients who were alive at the time of the database lock (March 31st, 2017) were administratively censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MLN9708
Number analyzed (Participants) | 12
months | NA [8.1 to NA] — The median overall survival time at 24 months could not be estimated. The lower bound of the 95% confidence interval was 8.1 months.

5. Secondary Outcome: Duration of Response
Description: Time from documentation of tumor response to disease progression.
Time Frame: 24 months after initiation of study treatment
Population: Although 12 patients were analyzable, only one patient responded to treatment and therefore only 1 patient is represented for the duration of response.
Measure: Number; unit: months
Arm/Group | MLN9708
Number analyzed (Participants) | 1
months | 12

ADVERSE EVENTS:
Arm/Group | MLN9708
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 8/12
Other Adverse Events (participants affected / at risk) | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MLN9708 (N=12)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Rash maculo-papular (Investigations) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MLN9708 (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes